CLINICAL TRIAL: NCT00002426
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Safety and Efficacy of Adefovir Dipivoxil as Intensification Therapy in Combination With Highly Active Antiretroviral Therapy (HAART) in HIV Infected Patients With HIV-1 RNA > 50 and <= 400 Copies/Ml
Brief Title: A Study on the Safety and Effectiveness of Adefovir Dipivoxil in Combination With Anti-HIV Therapy (HAART) in HIV-Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 232K; GS-97-415
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: HIV Infections
Keywords: HIV-1; RNA, Viral; VX 478; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil

SUMMARY:
The purpose of this study is to see if it is safe and effective to give an experimental anti-HIV drug, adefovir dipivoxil (ADV), in combination with other anti-HIV drugs (HAART) to patients who have a viral load (level of HIV in the blood) between 50 and 400 copies/ml.

DETAILED DESCRIPTION:
Patients are randomized to 1 of 2 arms in a 2:1 ratio. Approximately 260 patients receive ADV and approximately 130 patients receive placebo. Patients receive ADV or placebo in addition to L-carnitine and their current stable HAART regimen. Each patient receives blinded study medication for 48 weeks and is evaluated at Weeks 16, 24, and 48. Patients who reach the primary endpoint of virologic failure prior to Week 48 may continue blinded study medication or receive open-label ADV at the investigator's discretion. In both cases, patients continue their study visits as per the original visit schedule. Virologic failure is defined as 2 consecutive HIV-1 RNA measurements, after baseline, above 400 copies/ml (measured by the Roche Amplicor HIV-1 Monitor UltraSensitive assay) drawn at least 14 days apart. All patients who complete study visits without treatment-limiting ADV toxicity may continue open-label ADV in the Maintenance Phase at the discretion of the principal investigator.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have been on a stable HAART regimen consisting of at least 3 antiretroviral drugs for at least 16 weeks prior to study entry.
* Have a CD4 count of 50 cells/mm3 or more.
* Have a viral load greater than 50 and less than or equal to 400 copies/ml within 14 days prior to study entry.
* Have had at least 1 additional viral load in the past that was less than or equal to 400 copies/ml while on your current stable HAART regimen.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390

CONTACTS AND LOCATIONS:
Locations (49):
- United States (37):
  - Pacific Oaks Research, Beverly Hills, California
  - ViRx Inc, Palm Springs, California
  - Ctr for AIDS Research / Education and Service (CARES), Sacramento, California
  - San Francisco Gen Hosp / UCSF AIDS Program, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - San Francisco VA Med Ctr, San Francisco, California
  - Blick Med Associates, Stamford, Connecticut
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Dupont Circle Physicians Group, Washington D.C., District of Columbia
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - IDC Research Initiative, Altamonte Springs, Florida
  - Community AIDS Resource Inc, Coral Gables, Florida
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Duval County Health Department, Jacksonville, Florida
  - Health Positive, Safety Harbor, Florida
  - Center for Quality Care, Tampa, Florida
  - Georgia Research Associates, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana Univ Infectious Disease Research Clinic, Indianapolis, Indiana
  - Johns Hopkins Univ School of Medicine, Baltimore, Maryland
  - Albany Med College, Albany, New York
  - Bentley-Salick Med Practice, New York, New York
  - St Luke Roosevelt Hosp, New York, New York
  - James Jones MD, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Associates of Med and Mental Health, Tulsa, Oklahoma
  - The Research and Education Group, Portland, Oregon
  - Miriam Hosp, Providence, Rhode Island
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Vanderbilt Univ School of Medicine, Nashville, Tennessee
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Texas Med Branch, Galveston, Texas
  - Thomas Street Clinic, Houston, Texas
  - Univ of Utah Med School / Clinical Trials Ctr, Salt Lake City, Utah
  - Infectious Disease Physicians Inc, Annandale, Virginia
  - N Touch Research Corp, Seattle, Washington
- Canada (3):
  - St Paul's Hosp, Vancouver, British Columbia
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- France (2):
  - Hopital Edouard Herriot, Lyon
  - Hopital Sainte-Marguerite, Marseille
- Germany (3):
  - Klinikum Der Johann Wolfgang Goethe Universitat, Frankfurt
  - Universitatskrankenhaus Eppendorf, Hamburg
  - Klinikum der Ludwig-Maximilians-Universitaet, München
- United Kingdom (4):
  - Chelsea and Westminster Hosp, London
  - King's College Hospital, London
  - Royal Free Hosp, London
  - Senior Lecturer in GU Medicine, London